CLINICAL TRIAL: NCT06763146
Title: Real-world Experience With Finerenone Treatment in Patients From India With Chronic Kidney Disease and Type 2 Diabetes-Retrospective Data Analysis
Brief Title: An Observational Study to Learn More About How Safe Finerenone is and How Well it Works in Indian People With Chronic Kidney Disease and Type 2 Diabetes in Routine Medical Practice
Acronym: IN-REALITY
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22549
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes Mellitus
Keywords: CKD; T2DM
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Finerenone (Kerendia, BAY948862): Patients with CKD and T2D from India who initiate on finerenone per approved label.
  Interventions: Drug: Finerenone (Kerendia, BAY948862)

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY948862) — Retrospective cohort analysis using the investigator or a delegate at the study site collects secondary/historic data of finerenone usage (patient demographic and clinical characteristics, diagnosis-related, treatment-related, and laboratory data) from clinic specific medical records.

SUMMARY:
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.

Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

DETAILED DESCRIPTION:
This is an observational study in which data already collected from people with chronic kidney disease (CKD) and Type 2 diabetes mellitus (T2D) are studied.

T2D is a condition in which glucose levels rise in the blood. It is one of the common causes of CKD and can lead to kidney failure. CKD is a long-term condition in which the kidneys' ability to work properly gradually decreases over time.

The study drug, finerenone, is already approved for doctors to prescribe to people with CKD and T2D. It blocks the activity of a protein involved in worsening kidney function.

People with CKD and T2D are already receiving treatment with finerenone based on the results of previous studies. These studies, however, did not include Indian participants.

To better understand the impact of finerenone on CKD and T2D, more knowledge is needed about how well it works in the Indian population.

The main purpose of the study is to learn more about how well finerenone works and how safe it is in Indian people with CKD and T2D. To do this, researchers will check:

* participants' characteristics including age, sex, height and weight, and signs and symptoms of the disease
* other conditions the participants may have along with CKD and T2D, additional medicines they have taken with finerenone, and different treatment patterns in Indian participants.

The different treatment pattern for finerenone includes:

* specialty of the doctor who prescribed finerenone
* the date of starting finerenone
* whether participants were still taking finerenone at each follow-up visit
* the date and reason for stopping finerenone early
* the dose of finerenone the participants took and how often they took it
* changes in the dosage either with a low dose or high dose compared with the previous firenone dose
* after starting finerenone treatment: reseachers may ask to continue treatment with finerenone, or may suggest adding other treatments like SGLT2 inhibitors or potassium binders, or stop finerenone treatment
* after stopping finerenone treatment: researchers may start other treatments, like SGLT2 inhibitors, RAAS inhibitors, or potassium binders or other therapy

Researchers will only look at the medical records from participants in India. Data collected will be from August 2022 to April 2024.

Researchers will track participants' data in India and will follow them until the end of the study period till Nov 2024, last visit date of the participant, the participant discontinues treatment with finerenone, death, kidney failure, or cancer of the kidney.

In this study, only available data from routine care in India are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients from India (Indian ethnicity) diagnosed with CKD and T2D prior to initiating finerenone (per the standard diagnostic criteria) and initiated on finerenone per approved label.
* Patient was prescribed finerenone for the first time (drug naïve) for the management of CKD and T2D between 1st August 2022 and 30th April 2024.
* Age 18 years or older at the time of finerenone initiation.

Exclusion Criteria:

* eGFR <25 mL/min/1.73 m^2
* Serum potassium >5.0 mmol/L
* Type 1 diabetes is recorded in the patient record
* Contraindications according to the local marketing authorization - Patient data will be excluded if below information is identified in the patient record at any point from index date to the end of observation period:
* - Pregnancy.
* - Lactation.
* - Patient taking concomitant medications that are strong CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, ritonavir, nelfinavir, cobicistat, clarithromycin, telithromycin and nefazodone).
* - Addison's disease.
* Patient was a part of an interventional clinical study between 1st August 2022 and 30th Nov 2024.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of CKD associated with T2D who are initiated on finerenone under routine clinical management.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive summary of specialty of prescribing physician | Retrospective data analysis from 2022 to 2024
Date of finerenone initiation | Retrospective data analysis from 2022 to 2024
If patient was receiving finerenone at the time of each follow-up visit (Yes/No) | Retrospective data analysis from 2022 to 2024
Date of discontinuation of finerenone | Retrospective data analysis from 2022 to 2024
Reason for discontinuation of finerenone | Retrospective data analysis from 2022 to 2024
Dose of finerenone treatment | Retrospective data analysis from 2022 to 2024
Frequency of finerenone treatment | Retrospective data analysis from 2022 to 2024
The number of patients who initiated finerenone with a 10-mg dose and 20-mg dose | Retrospective data analysis from 2022 to 2024
The proportion of patients who initiated finerenone with a 10-mg dose and have up-titrated to a 20-mg dose | Retrospective data analysis from 2022 to 2024
The proportion of patients who initiated finerenone with a 20-mg dose and have down-titrated to a 10-mg dose | Retrospective data analysis from 2022 to 2024
Actions taken after finerenone introduction | Retrospective data analysis from 2022 to 2024
  Actions include continue treatment, addition of second therapy like SGLT2is, potassium binders, discontinue treatment
Actions taken after stop finerenone prescription | Retrospective data analysis from 2022 to 2024
  Actions include initiate alternate therapy like Sodium-glucose transport protein-2 inhibitor (SGLT2is), RAASis or potassium binders, other

SECONDARY OUTCOMES:
UACR (mg/g) before and after initiating finerenone | Retrospective data analysis from Aug 2022 to Apr 2024
  UACR: Urine Albumin to Creatinine Ratio
eGFR before and after initiating finerenone | Retrospective data analysis from Aug 2022 to Apr 2024
  eGFR: Estimated glomerular filtration rate
Serum potassium (mmol/L) before and after initiating finerenone | Retrospective data analysis from Aug 2022 to Apr 2024
Change in UACR after initiating finerenone vs month 1, month 4 and end of study | Retrospective data analysis from 2022 to 2024
Change in serum potassium after initiating finerenone vs month 1, month 4 and end of study | Retrospective data analysis from Aug 2022 to Apr 2024
Change in Serum creatinine/eGFR after initiating finerenone vs month 1, month 4 and end of study | Retrospective data analysis from Aug 2022 to Apr 2024
Frequency of events like hospitalization and dialysis due to hyperkalemia | Retrospective data analysis from Aug 2022 to Apr 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, India

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.